CLINICAL TRIAL: NCT00371397
Title: Psychoneuroimmunology and Mind-Body Interventions
Brief Title: Yoga, Immune Function, and Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Janice Kiecolt-Glaser, Director, Institute for Behavioral Medicine Research, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2005H0068; R21AT002971-01 (NIH)
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2011-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: yoga; immune function; stress; health; mood; skin barrier repair

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hatha yoga classes (Experimental): Groups consisted of novices or experts. Groups were counterbalanced to ensure that equal number of novices and experts participated in each possible session combination, in a randomly assigned order.
  Interventions: Behavioral: Hatha Yoga Classes
- Movement Control (Sham Comparator): Non-Hatha yoga gentle movement. Groups consisted of novices or experts. Groups were counterbalanced to ensure that equal number of novices and experts participated in each possible session combination, in a randomly assigned order.
  Interventions: Behavioral: Movement Control
- Passive Video Control (No Intervention): Another control condition, a neutral video that did not include any music, allowed us to contrast the effects of yoga with no activity.The session included a sequence on how to design physics experiments for a high school classroom, as well as segments from two lectures on polymers and quantum mechanics. Groups were counterbalanced to ensure that equal number of novices and experts participated in each possible session combination, in a randomly assigned order.

INTERVENTIONS:
Behavioral: Hatha Yoga Classes — Iyengar yoga, the form of hatha yoga used in this study, emphasizes the use of props to help students achieve precise postures safely and comfortably according to their particular body types and needs. The yoga activity sessions were directed by four experienced yoga teachers following a script. The poses used were (in order) Supta Baddha Konasana (Reclining Bound Angle Pose), Adho Mukha Svanasana (Downward Facing Dog), Supported Uttanasana (Intense Forward Stretch), Parsvotanasana (Intense Side Stretch Pose), Prasarita Padottanansana (Wide-Legged Forward Bend), Janu Sirsasana (Head to Knee Pose), Bharadvajasana (Simple Seated Twist Pose), Viparita Karani (Restful Inversion), Supported Setu Bandha Sarvanagasana (Bridge Pose), and Savasana (Corpse Pose). Blood draws occurred during the last two minutes of Supta Baddha Konasana (pose held 10 minutes), Viparita Karani (10 minutes), and Savasana (15 minutes).
  Arms: Hatha yoga classes
Behavioral: Movement Control — Walking on a treadmill at .5 miles per hour was used to control for general physical movement/cardiovascular expenditure because it best approximated the heart rates during the restorative yoga session. To match the lower heart rate, women also rested supine on a bed for several minutes after walking, before and after getting their blood drawn.
  Arms: Movement Control

SUMMARY:
This study is designed to examine the impact of hatha yoga on immune and hormonal functioning in healthy individuals.

DETAILED DESCRIPTION:
This study is designed to examine the effects of hatha yoga on autonomic, immune, and endocrine function. The data from both inexperienced and experienced groups will help us better understand how longer-term practice of yoga may be beneficial. The study consists of one 3-hour screening session and three 6-hour activity sessions with 30 minute follow-up appointments the following morning scheduled 2 - 4 weeks apart. Each participant will complete the 3 activity sessions, which will consist of either yoga, mild movement, or a neutral activity (watching a videotape), in randomly assigned order. Thus, both novices and experts will participate in 3 activity sessions each (yoga, movement control, video control). The order in which each participant goes through the activity sessions is counterbalanced. Data for each activity session will be aggregated by group (i.e. novice or expert). We will measure responses to tape stripping to assess skin barrier repair, and evaluate responses to computer tasks, self-report measures, and a battery of unobtrusive behavioral measures. We will also collect blood and saliva samples to measure immune and endocrine outcomes.

ELIGIBILITY:
Inclusion Criteria:

* healthy female adults
* relatively inexperienced with yoga (beginner)
* experienced with yoga (advanced practitioner)

Exclusion Criteria:

* Treatment with medication that has immunological or endocrinological consequences
* Chronic health problems that affect immune or endocrine systems
* Anemia
* Use of psychoactive drugs or mood-altering medication
* Smoking
* Needle or blood phobias
* Tape or bandage allergies
* Pregnancy or nursing within the previous 3 months
* Heart problems
* History of hip or knee replacement surgery, displaced vertebrae, and any other physical limitations that would prevent full participation in the program
* use of statins, beta blockers
* excessive alcohol use
* convulsive disorders
* Body Mass Index (BMI) ≥ 30.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice K. Kiecolt-Glaser, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Clinical Research Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Kiecolt-Glaser JK, Christian L, Preston H, Houts CR, Malarkey WB, Emery CF, Glaser R. Stress, inflammation, and yoga practice. Psychosom Med. 2010 Feb;72(2):113-21. doi: 10.1097/PSY.0b013e3181cb9377. Epub 2010 Jan 11. PMID 20064902
- See also: Please click here to visit our website if you would like to read more about our studies. — http://www.stressandhealth.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited through online ads and notices posted in yoga studios. All women participated in some form of hatha yoga.
Groups:
- Expert: Movement Control Then Hatha Yoga Then Video: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Hatha Yoga Class in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning.
- Expert: Hatha Yoga Then Video Then Movement Control: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Hatha Yoga Class in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning.
- Expert: Video Then Movement Control Then Hatha Yoga: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Hatha Yoga Class in 1 day and a 30 minute follow-up session the next morning.
- Expert: Movement Control Then Video Then Hatha Yoga: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Hatha Yoga session in 1 day and a 30 minute follow-up session the next morning.
- Expert: Hatha Yoga Then Movement Control Then Video: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning.
- Expert: Video Then Hatha Yoga Then Movement Control: Participants are female Yoga experts, meaning they have practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
  * For Session 1, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Movement Control Activity in 1 day and a 30 minute follow-up session the next morning.
- Novice: Movement Control Then Hatha Yoga Then Video: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning.
- Novice: Hatha Yoga Then Video Then Movement Control: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning.
- Novice: Video Then Movement Control Then Hatha Yoga: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Hatha Yoga session in 1 day and a 30 minute follow-up session the next morning.
- Novice: Movement Control Then Video Then Hatha Yoga: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Movement Control Activity in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Hatha Yoga session in 1 day and a 30 minute follow-up session the next morning.
- Novice: Hatha Yoga Then Movement Control Then Video: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Movement Control Activity in 1 day and a 30 minute follow-up session the next morning.
  * For Session 3, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
- Novice: Video Then Hatha Yoga Then Movement Control: Participants are female Yoga novices, meaning they had participated in yoga classes or practiced at home with yoga videos for 6 - 12 sessions.
  * For Session 1, participants completed the Video Control Activity in 1 day and a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 2, participants completed the Hatha Yoga session in 1 day, a 30 minute follow-up session the next morning, followed by 2-4 weeks of normal daily activity.
  * For Session 3, participants completed the Movement Control Activity in 1 day and a 30 minute follow-up session the next morning.
Period: Session 1
Arm/Group | Expert: Movement Control Then Hatha Yoga Then Video | Expert: Hatha Yoga Then Video Then Movement Control | Expert: Video Then Movement Control Then Hatha Yoga | Expert: Movement Control Then Video Then Hatha Yoga | Expert: Hatha Yoga Then Movement Control Then Video | Expert: Video Then Hatha Yoga Then Movement Control | Novice: Movement Control Then Hatha Yoga Then Video | Novice: Hatha Yoga Then Video Then Movement Control | Novice: Video Then Movement Control Then Hatha Yoga | Novice: Movement Control Then Video Then Hatha Yoga | Novice: Hatha Yoga Then Movement Control Then Video | Novice: Video Then Hatha Yoga Then Movement Control
Started | 5 | 7 | 5 | 2 | 3 | 4 | 4 | 5 | 6 | 5 | 4 | 2
Completed | 4 | 7 | 5 | 2 | 3 | 4 | 4 | 4 | 6 | 5 | 4 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Session 2
Arm/Group | Expert: Movement Control Then Hatha Yoga Then Video | Expert: Hatha Yoga Then Video Then Movement Control | Expert: Video Then Movement Control Then Hatha Yoga | Expert: Movement Control Then Video Then Hatha Yoga | Expert: Hatha Yoga Then Movement Control Then Video | Expert: Video Then Hatha Yoga Then Movement Control | Novice: Movement Control Then Hatha Yoga Then Video | Novice: Hatha Yoga Then Video Then Movement Control | Novice: Video Then Movement Control Then Hatha Yoga | Novice: Movement Control Then Video Then Hatha Yoga | Novice: Hatha Yoga Then Movement Control Then Video | Novice: Video Then Hatha Yoga Then Movement Control
Started | 4 | 7 | 5 | 2 | 3 | 4 | 4 | 4 | 6 | 5 | 4 | 2
Completed | 4 | 7 | 5 | 2 | 3 | 4 | 4 | 4 | 6 | 5 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Session 3
Arm/Group | Expert: Movement Control Then Hatha Yoga Then Video | Expert: Hatha Yoga Then Video Then Movement Control | Expert: Video Then Movement Control Then Hatha Yoga | Expert: Movement Control Then Video Then Hatha Yoga | Expert: Hatha Yoga Then Movement Control Then Video | Expert: Video Then Hatha Yoga Then Movement Control | Novice: Movement Control Then Hatha Yoga Then Video | Novice: Hatha Yoga Then Video Then Movement Control | Novice: Video Then Movement Control Then Hatha Yoga | Novice: Movement Control Then Video Then Hatha Yoga | Novice: Hatha Yoga Then Movement Control Then Video | Novice: Video Then Hatha Yoga Then Movement Control
Started | 4 | 7 | 5 | 2 | 3 | 4 | 4 | 4 | 6 | 5 | 4 | 2
Completed | 4 | 7 | 5 | 2 | 3 | 4 | 4 | 4 | 6 | 5 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Women were exposed to each of the conditions (yoga, movement control, and passive-video control) during three separate visits. The order of the visits was randomized per participant. 52 total participants enrolled.
Arm/Group | Overall Study
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.32 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detectable C-Reactive Protein (CRP)
Description: High sensitivity C-reactive protein (hsCRP) assessed once at baseline, at each of the three visits. The hsCRP assay was performed using chemiluminescence methodology with the Immulite 1000 (Siemens Medical Solutions, Los Angeles, Ca.) The lowest level of detection is .3 mg/dL. 43% of the values were below this lower bound, thus hsCRP was dichotomized as undetectable/detectable.
Time Frame: 8:30 a.m. at each of the three visits, scheduled at least 2 weeks apart
Measure: Number; unit: participants with CRP above 0.3
Groups:
- Novice: Women were classified as novices if they had participated in yoga classes or home practice with yoga videos for 6 - 12 sessions.
- Expert: Women were classified as Experts if they had practiced yoga regularly 1-2 times per week (75-90 min sessions) for at least 2 years, and at least 2 times per week for the past year.
Arm/Group | Novice | Expert
Number analyzed (Participants) | 25 | 25
participants with CRP above 0.3 | 16 | 8
Statistical Analysis 1: Comparison: Novice vs Expert; hsCRP dichotomized as undetectable/detectable. Logistic regression w/generalized estimating equations(GEE)s to determine odds ratio. Assessed hsCRP at baseline at each of the three visits; 43% of the values (n = 65) were below the assay's detectable lower bound of .3 mg/dL, and thus hsCRP was dichotomized as undetectable/detectable; Test type: Superiority or Other; p = .009, Regression, Logistic; Odds Ratio (OR) = 4.75

2. Primary Outcome: Cortisol
Description: All cortisol and catecholamine samples for a subject were frozen after collection and analyzed within the same assay run after the participant had completed the study.
Time Frame: Day 1 8:30, 10:05, 10:58, 11:35, 12:05, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: pg/ml

3. Primary Outcome: Skin Barrier Repair: Trans-epidermal Water Loss (TEWL)
Description: Cellophane tape stripping, a common dermatological paradigm for studying restoration of the skin barrier, was used to examine whether the time necessary for recovery from minor physical insults varied by condition or yoga expertise. Measurement of the rate of transepidermal water loss (TEWL) through human skin provides a noninvasive method to monitor changes in the skin's barrier function. TEWL was measured twice during the session using a computerized evaporimetry instrument, the DermaLab® (CyberDERM, Media, PA), and barrier recovery was calculated.
Time Frame: 11:50, 12:50 at each of the three visits, scheduled at least 2 weeks apart
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: number tape strips

4. Primary Outcome: Immune Function: Soluble Interleukin-6 Receptor (sIL-6r)
Description: Serum levels of the sIL-6r were assayed using Quantikine High Sensitivity Immunoassay kits (R&D), per kit instructions.
Time Frame: Day 1 8:30, 11:35, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml

5. Primary Outcome: Immune Function: Tumor Necrosis Factor-alpha (TNF-α)
Description: Serum levels of TNF-α were assayed using Quantikine High Sensitivity Immunoassay kits (R&D), per kit instructions.
Time Frame: Day 1 8:30, 11:35, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml (log 10)

6. Primary Outcome: Immune Function: Lipopolysaccharide (LPS) -Stimulated Production of Interleukin-6 (IL-6)
Description: Supernatants from PBLs stimulated with 5μg/ml lipopolysaccharide (LPS) for 72 h were assayed for IL-6 and TNF-α using ELISA kits (B-D Pharmingen).
Time Frame: Day 1 8:30, 10:05, 11:35, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml

7. Primary Outcome: Immune Function: LPS-stimulated Production of TNF-α
Description: as for outcome 6
Time Frame: Day 1 8:30, 10:05, 11:35, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml

8. Primary Outcome: Immune Function: Interleukin-6 (IL-6)
Description: Serum levels of TNF-α, IL-6, and the sIL-6r were assayed using Quantikine High Sensitivity Immunoassay kits (R&D), per kit instructions
Time Frame: Day 1 8:30, 11:35, 13:10. Day 2 7:30
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml (log 10)

9. Primary Outcome: Catecholamine Production: Epinephrine
Description: as for outcome 2
Time Frame: 8:30, 10:05, 10:28, 10:58, 11:35, 12:05 at each of the three visits, scheduled at least 2 weeks apart
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml (log 10)

10. Primary Outcome: Catecholamine Production: Norepinephrine
Description: as for outcome 2
Time Frame: 8:30, 10:05, 10:28, 10:58, 11:35, 12:05
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pg/ml (log 10)

11. Secondary Outcome: Heart Rate
Time Frame: Day 1: 8:30, 9:15, 9:45, 10:00, 10:45, 11:35, 12:05, 12:15
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: bpm

12. Secondary Outcome: Blood Pressure
Time Frame: 7:55 at each of the three visits, scheduled at least 2 weeks apart
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mmHg

13. Secondary Outcome: Mood: Positive and Negative Affect Schedule (PANAS)Positive
Description: The Positive and Negative Affect Schedule (PANAS) includes two 10-item mood scales. Each item is rated on a 5-point scale ranging from 1 = very slightly or not at all to 5 = extremely, to indicate the extent to which the respondent has felt this way in the indicated time frame. Several additional words were added to better capture low positive affect: happy, satisfied, disappointed, discouraged, low, sad.
Time Frame: 7:35, 11:45, 12:30 at each of the three visits, scheduled at least 2 weeks apart
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Cumulative Score, 0-50

14. Secondary Outcome: Mood: Positive and Negative Affect Schedule (PANAS)Negative
Description: as for outcome 13
Time Frame: 7:35, 11:45, 12:30 at each of the three visits, scheduled at least 2 weeks apart
Reporting Status: Not Posted
Measure: Number; unit: Cumulative Score, 0-50

ADVERSE EVENTS:
Arm/Group | Novice | Expert
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes